CLINICAL TRIAL: NCT06250179
Title: 3D VOLUMETRIC CHANGE OF THE PALATAL DONOR REGION IN WOUND HEALING
Acronym: (DIMENSIONAL)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Collaborators: DİLEK ÖZKAN ŞEN (Unknown)
Responsible Party: Principal Investigator, FATMA SARAÇ, research assistant, Necmettin Erbakan University
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Screening
Other Study IDs: necmettinerbakanü
Record Dates: First submitted 2024-02-01; First posted 2024-02-08 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Free Gingival Graft Volume Change
Keywords: free gingival graft; cigarette; 3D scanning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-smoking patients (Experimental): The patient will receive a free gingival graft for insufficient keratinized gingival height.
  Interventions: Procedure: free gingiva graft surgery
- 'Light' smokers who report smoking less than 5 cigarettes per day (Active Comparator): The patient will receive a free gingival graft for insufficient keratinized gingival height.
  Interventions: Procedure: free gingiva graft surgery
- Non-smoker for 5 years, quit smoking patients (Active Comparator): The patient will receive a free gingival graft for insufficient keratinized gingival height.
  Interventions: Procedure: free gingiva graft surgery

INTERVENTIONS:
Procedure: free gingiva graft surgery — For insufficient gingival height in patients, the free gingival graft taken from the palate will be sutured to the relevant area.

SUMMARY:
The purpose of this clinical trial is planned to be conducted with 45 individuals aged between 18-65, with Cairo type I gingival recession and patients requiring free gingival surgery. It was aimed to investigate when the palatal mucosa will return to its previous volume in the donor area and the effect of smoking. The main questions it aims to answer are:

* Evaluation of 3D volume change of the palatal donor area from which free gingival graft was taken
* determining how long it takes for the palatal mucosa to regain its original shape and thickness Participants will be asked to comply with postoperative recommendations and pay attention to oral hygiene.

If there is a comparison group: Researchers use it to see if smoking affects the volume change in the donor area.

They will compare non-smokers with clinically healthy gums, 'light' smokers who report smoking less than 5 cigarettes per day and patients with clinically healthy gums, and ex-smokers with clinically healthy gums who have not smoked for 5 years.

DETAILED DESCRIPTION:
This study is planned to be conducted with 45 individuals aged between 18-65 who applied to Necmettin Erbakan University Faculty of Dentistry Department of Periodontology for various reasons. In the Department of Periodontology, each patient diagnosed with periodontal disease after clinical and radiological evaluation is initially treated with phase-1 treatment. In addition, the treatment of patients with mucogingival problems (gingival recession, keratinized gingival insufficiency, shallow vestibule depth) whose phase-1 treatment has been completed in our periodontology clinic continues (with free gingival graft and connective tissue graft surgery, etc.). Pre- and post-operative clinical measurements and photographs of patients for whom surgical procedures are planned are taken and kept in our archive.

In this prospectively planned study, the palatal area of patients who have received an indication for free gingival surgery for any reason and who meet the inclusion criteria and have agreed to participate in the study will be scanned with an intraoral scanner before and after the procedure, and the changes in palate volume will be monitored at 1st and 3rd month follow-ups.

Inclusion and exclusion criteria (limitations):

Study inclusion criteria:

1. Volunteers aged 18 and over
2. Patients with Cairo type I gingival recession and requiring free gingival surgery
3. Not having a psychiatric, mental or physical disability
4. Not having received periodontal treatment in the last 6 months
5. Being systemically healthy
6. Having at least 20 teeth in your entire mouth
7. Getting diagnosed with healthy gums
8. Not using any medication
9. Not being pregnant
10. Not having used any antibiotics, anti-inflammatory or any other drugs that may affect periodontal tissues in the last 6 months for any reason.

Exclusion criteria from the study:

1) Being outside the inclusion criteria and not agreeing to participate in the study individual selection If the patients who come to the Periodontology Clinic Secretariat for periodontal treatment meet the inclusion criteria of the study whose Phase-1 treatment has been completed, the patients who accept the study and those who sign the consent form will be included in the study.

Considering the possibility of participants dropping out of the study, the number of individuals to be included in each group was determined as 15 and it is planned to be conducted with 45 individuals in total.

Group 1: Patients who are non-smokers and have clinically healthy gums Group 2: 'Light' smokers who report smoking less than 5 cigarettes per day and patients with clinically healthy gums Group 3: Patients with clinically healthy gums and ex-smokers who have not smoked for 5 years.

An intraoral optical scanner (TRIOS, 3Shape) will be used to obtain digital models as STL files at baseline (before surgery) and at 1 and 3 months. STL files will be imported into a digital imaging software (Geomagic Control X®) to measure donor site volume changes over time. All digital volumetric analyzes will be performed. STL files from baseline and follow-up visits will be overlaid and matched using the most appropriate algorithm. Stable anatomical landmarks (teeth and contralateral palate) will be used to perform overlay of models to guarantee maximum accuracy of digital analysis. Observed volumetric results are planned to include: average volumetric (Volume) changes, average distance between surfaces (difference in average thickness of the reconstructed volume; DD), and linear dimensional changes (LD) at points 3, 5, and 7 mm. Patient age, gender, and graft dimensions (width, height, and thickness) will also be recorded. The primary outcome of this study is to observe the post-operative dimensional changes of donor areas at different follow-up periods by evaluating them in volumetric and linear dimensions. The secondary outcome is to evaluate volumetric outcomes (such as gender, age, and graft size) together with patient (including smoking) and surgery-related factors that may affect the outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers aged 18 and over
2. Treatments with Cairo type I gingival treatment and requiring free gingival surgery
3. There is no psychiatric, mental or physical disability
4. My son has not received periodontal treatment within 6 months.
5. Being systemically healthy
6. Having at least 20 teeth in your entire mouth
7. Getting diagnosed with healthy gums
8. Not using any medication
9. Not pregnant
10. Not having used any antibiotics, anti-inflammatory or any other medication that will swell the periodontal tissues in the last 6 months for any reason.

Exclusion Criteria:

1) Being outside the inclusion criteria and not agreeing to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Examination of volume change in the palatal donor region in smoking and non-smoking patients | 3 months
  It was aimed to examine the volume change among the 3 groups in our study by looking at its connection with smoking. A study plan was created by comparing the 3D shape device on which the scans were made with Geomatic Control X and looking at the volume change.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan Üniversitesi, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Free gingiva in non-smoking patients with insufficient keratinized gingival height and clinically healthy gingiva, 'light' smokers who report smoking less than 5 cigarettes per day and patients with clinically healthy gingiva, and patients with healthy gingiva who have quit smoking and have not smoked for 5 years. It was aimed to evaluate the 3D volume change of the grafted palatal donor area, to determine the volumetric change in the donor area and how long it took for the palatal mucosa to regain its original shape and thickness.
Supporting Information: Study Protocol, SAP
Time Frame: February 2024-July 2024
Access Criteria: search